CLINICAL TRIAL: NCT04854135
Title: Continuous Glucose Monitoring Initiation at Hospital Discharge: A Feasibility Pilot Study
Brief Title: Continuous Glucose Monitoring Initiation at Hospital Discharge
Acronym: CGM4Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High drop out rate
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Paulina Cruz Bravo, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202101175
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes; Type2 Diabetes; Hyperglycemia; Hypoglycemia; Hypoglycemia Unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CGM Intervention (Experimental): All eligible patients will receive a Continuous Glucose Monitor (CGM) prior to hospital discharge after signing an informed consent.
  Interventions: Device: CGM4Home

INTERVENTIONS:
Device: CGM4Home — FreeStyle Libre 2 Continuous Glucose Monitoring System manufactured by Abbott

SUMMARY:
The purpose of this study is to look at feasibility (the likelihood) of continued use of the FreeStyle Libre 2 Continuous glucose monitor (CGM) when started at the time of hospital discharge in patients with poorly controlled diabetes and to look at the effects of CGM use on blood glucose control and quality of life. Additional information will be collected to determine the barriers to continuing CGM use after discharge. The investigators will also collect information to see how well blood glucose has been controlled after discharge while utilizing the CGM.

DETAILED DESCRIPTION:
VISIT/PHONE CALL WHAT WILL HAPPEN? (estimated time) [window]

Screening Visit (~45 minutes) Review consent form and obtain consent Complete questionnaire, obtain diabetes history Day of Discharge (~1 hour) Complete FreeStyle Libre 2 CGM education Attach FreeStyle Libre 2 CGM sensor to arm Within 1-3 weeks from discharge Phone Call (~30 minutes) Questions regarding use of FreeStyle Libre 2 CGM Current diabetes regimen Adverse Events Reminder to take FreeStyle Libre 2 CGM sensor prescription to pharmacy to be filled

1 & 3 Month Phone Call (~45 minutes) [+/- 5 days] Questions regarding use of FreeStyle Libre 2 CGM Current diabetes regimen Complete questionnaire Adverse Events 6 Month Phone Call (~15 minutes) [+/- 10 days] Questions regarding use of FreeStyle Libre 2 CGM Barriers to FreeStyle Libre 2 CGM use

Validated Instruments: Diabetes self-management Questionnaire (DMSQ)

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Have diabetes (type 1 diabetes mellitus, type 2 diabetes mellitus, cystic fibrosis related diabetes mellitus)
3. Hemoglobin A1c greater than or equal to 8.0% or history of hypoglycemia unawareness
4. Able and willing to sign informed consent form
5. Have a valid telephone number
6. Willing to purchase FreeStyle Libre 2 CGM sensors out of pocket after discharge from hospital (when insurance coverage isn't available)

Exclusion Criteria:

1. Unable to sign informed consent form
2. Have altered mental status
3. Unable to manage diabetes independently at home
4. Have utilized CGM in the past
5. Pregnancy
6. New steroid-induced hyperglycemia
7. Unwilling to participate in the study
8. Have kidney disease requiring hemodialysis
9. Taking high doses of vitamin C daily (greater than 500 mg every day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Cruz Bravo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital/ Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graber AL, Davidson FA, Brown MS, Gaume JA, McRae MD, Wolff K. Hospitalization of patients with diabetes. Endocr Pract. 1995 Nov-Dec;1(6):399-403. doi: 10.4158/EP.1.6.399. PMID 15251567
- [Background] Mattishent K, Lane K, Salter C, Dhatariya K, May HM, Neupane S, Loke YK. Continuous glucose monitoring in older people with diabetes and memory problems: a mixed-methods feasibility study in the UK. BMJ Open. 2019 Nov 18;9(11):e032037. doi: 10.1136/bmjopen-2019-032037. PMID 31740472
- [Background] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Background] Beck RW, Riddlesworth TD, Ruedy K, Ahmann A, Haller S, Kruger D, McGill JB, Polonsky W, Price D, Aronoff S, Aronson R, Toschi E, Kollman C, Bergenstal R; DIAMOND Study Group. Continuous Glucose Monitoring Versus Usual Care in Patients With Type 2 Diabetes Receiving Multiple Daily Insulin Injections: A Randomized Trial. Ann Intern Med. 2017 Sep 19;167(6):365-374. doi: 10.7326/M16-2855. Epub 2017 Aug 22. PMID 28828487
- [Background] Ehrhardt NM, Chellappa M, Walker MS, Fonda SJ, Vigersky RA. The effect of real-time continuous glucose monitoring on glycemic control in patients with type 2 diabetes mellitus. J Diabetes Sci Technol. 2011 May 1;5(3):668-75. doi: 10.1177/193229681100500320. PMID 21722581
- [Background] Yoo HJ, An HG, Park SY, Ryu OH, Kim HY, Seo JA, Hong EG, Shin DH, Kim YH, Kim SG, Choi KM, Park IB, Yu JM, Baik SH. Use of a real time continuous glucose monitoring system as a motivational device for poorly controlled type 2 diabetes. Diabetes Res Clin Pract. 2008 Oct;82(1):73-9. doi: 10.1016/j.diabres.2008.06.015. Epub 2008 Aug 12. PMID 18701183
- [Background] Whelan ME, Orme MW, Kingsnorth AP, Sherar LB, Denton FL, Esliger DW. Examining the Use of Glucose and Physical Activity Self-Monitoring Technologies in Individuals at Moderate to High Risk of Developing Type 2 Diabetes: Randomized Trial. JMIR Mhealth Uhealth. 2019 Oct 28;7(10):e14195. doi: 10.2196/14195. PMID 31661077

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGM Intervention
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CGM Intervention
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Black Non Hispanic White Non Hispanic Hispanic/Latino
  Participants
    Black Non Hispanic | 9
    White, Non Hispanic | 10
    Hispanic/Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Feasibility of Initiating a Continuous Glucose Monitoring in Patients With Diabetes at Hospital Discharge
Description: Starting and continuing to use a CGM at this critical time is feasible. Feasibility is defined as at least 20 percent of patients with diabetes referred for diabetes education meet inclusion criteria to participate and at least 75 percent participate. From those who participate, at least 50 percent continue using the CGM at 3 months.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Intervention
Number analyzed (Participants) | 20
Participants
  Lost to follow up | 13
  Discontinued use at 3 months | 3
  Continued use at 3 months | 4

2. Secondary Outcome: Percentage of Patients That Discontinue the CGM
Description: Discontinuation rate, measured by percentage of patients that discontinue the CGM at 6 months with wearing device, use, costs, getting refills, etc.)
Time Frame: At 6 months
Population: Participants lost to follow up were counted as discontinued
Measure: Count of Participants; unit: Participants
Groups:
- Discontinued Use: at 6 months
Arm/Group | Discontinued Use
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Mean Time in Range Outcomes
Description: Mean and SD of Time below target, in target and above target at 1 month and 3 months
Time Frame: At 1 month and 3 months
Population: Data was not collected
Arm/Group | CGM Intervention
Number analyzed (Participants) | 0

4. Secondary Outcome: Mean Change in Self-efficacy at 3 Months
Description: Using the Diabetes self-management Questionnaire (DMSQ), the investigators will measure the mean change and SD in the score (pre- and post- intervention)
  score is 0-48, higher scores mean a better outcome
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CGM Intervention Baseline; 3-month: All eligible patients will receive a Continuous Glucose Monitor (CGM) prior to hospital discharge after signing an informed consent.
  CGM4Home: FreeStyle Libre 2 Continuous Glucose Monitoring System manufactured by Abbott
Arm/Group | CGM Intervention Baseline | 3-month
Number analyzed (Participants) | 12 | 5
score on a scale | 30.66 (8.2) | 40.8 (7.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CGM Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT04854135/Prot_SAP_001.pdf